CLINICAL TRIAL: NCT02348346
Title: Effect of MVX (Titanium Dioxide) on the Microbial Colonization of Surfaces in an Intensive Care Unit
Acronym: TITANIC
Status: Completed | Type: Observational
Sponsor: drs. B. de Jong (Other)
Responsible Party: Sponsor-Investigator, drs. B. de Jong, MD, Gelderse Vallei Hospital
Organization: Gelderse Vallei Hospital (Other)
Other Study IDs: MVX 1.0
Record Dates: First submitted 2015-01-15; First posted 2015-01-28 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Environmental Contamination
Keywords: self-disinfecting surfaces; titanium dioxide
MeSH Terms: interventions — titanium dioxide

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: MVX (titanium dioxide) — The investigators have designed a prospective pre-post evaluation time-based pilot study addressing the microbial colonization of surfaces in four rooms of the ICU before and after coating with titanium dioxide (MVX). During a pre-intervention period cultures will be taken every 7 days from 10 prespecified and marked sites per room for a total duration of 4 weeks (sink, wall, floor, bed rail, door handle, ceiling, keyboard patient room, nurse call button, bedside table and monitor arm). After coating of the rooms with MVX another 4 weeks observation period will be used to gather samples in the post-intervention period.

SUMMARY:
Environmental cleanliness As antimicrobial resistance is a major and overall deteriorating public health problem international cooperation is necessary. Continued progress is needed to implement and improve programmes for the prevention and control of antimicrobial resistance and HAIs.

Environmental cleanliness might be one of the most important initiatives to reduce HAIs. Hospital surfaces are heavily contaminated with bacteria with the highest numbers on surfaces closest to the patients. Bed rails, nurse call buttons, curtains, towel dispensers, door handles, sinks, floors, clinical information stations, medical devices, stethoscopes, staff toilets etc. Actually, general hospital wards and Intensive Care Units are loaded with an abundance of potential pathogens 8,9,10. Surviving days, weeks or even months in the environment 11. Colonizing patients with bacteria from the hospital environment and getting HAIs or even die.

As most ventilator-associated pneumonias (VAPs) are the result of nosocomial microorganisms the environment plays an important role in the acquisition of pathogenic bacteria by contaminating health care workers hands and equipment 12,13. Furthermore, ICUs and wards struggle with colonized patients with ESBL-bacteria from sinks eventually leading to dead or outbreaks of group A streptococcus infections from contaminated curtains 14,15.

As key healthcare-associated pathogens have the capacity to persist for weeks to months on hospital surfaces indirect transmission is a serious threat, especially as antimicrobial resistance increases. Hospitalization in a room in which the previous patient had been colonized or infected with nosocomial pathogens (e.g. MRSA, VRE, multidrug-resistant Acinetobacter, Pseudomonas or C. difficile) has been shown to be a risk factor for colonization of infection with the same pathogen for the next patient16. Furthermore, the most important risk factor for hand and glove contamination of healthcare workers with multidrug-resistant bacteria has been demonstrated to be positive environmental cultures 17. To decrease the frequency and level of contamination of environmental surfaces the Centre for Disease Control and Prevention recommends routine disinfection of medical equipment and environmental surfaces to prevent the spread of potential pathogens through the hospital ward or ICU 18. Improved room cleaning has shown to decrease the risk for MRSA, VRE and C. difficile acquisition. Unfortunately, environmental cleaning is frequently inadequate. Less than 50% of hospital room surfaces are adequately cleaned and disinfected even by environmental services personnel. Environmental services personnel have low wages, are under time pressure to clean rooms quickly with high turn-over rates of patients. Novel materials and cleaning technologies have been developed as ultraviolet germicidal irradiation (UVGI) or hydrogen peroxide vapor (HPV). However, both technologies are expensive and can just be used for terminal cleaning and not during routine daily care 16. Self-disinfecting surfaces may overcome these problems. Once applied antimicrobial surfaces will continuously reduce the bioburden of nosocomial pathogens preventing transmission and decrease HAIs.

MVX One of these self-disinfecting products is MVX. MVX contains titanium dioxide which by the use of nanotechnology is now available for use in the health sector. Working as a photocatalyticum it generates, in the presence of light, hydroxy radicals and oxygen radicals for at least five years after coating hospital surfaces (durability test TUV Rheinland). Laboratory tests show that MVX is effective in killing bacteria, viruses and fungi (see attachment 1 for summary test results).

The positive results reported on the effects of MVX from laboratory evaluations still have to be confirmed in the clinical setting. After getting the CE-marking Gelderse Vallei Hospital in Ede, the Netherlands, will be the first hospital in Europe to study the efficacy of MVX in the Intensive Care Unit (ICU).

DETAILED DESCRIPTION:
Introduction and background

Background The annual epidemiological report and annual report of the EARS-NET of the European Centre for Disease Prevention and Control (ECDC) describes a continuing deteriorating situation in European countries. Antimicrobial resistance is increasing in Escherichia coli and Klebsiella pneumoniae isolates and surveillance data show high percentages of ESBL-positive isolates. Of particular concern is the increased percentage of Klebsiella pneumoniae and other bacterial groups resistant to carbapanems (last line antibiotics). Furthermore, the percentage of methicillin-resistant Staphylococcus aureus is still high and remains a public health priority On any given day 5.7% of the patients in European hospitals has a healthcare-associated infection (HAI) with a prevalence of at least one HAI of 19.5% for patients admitted to Intensive Care Units. HAIs are accountable for at least 37000 attributable deaths with annual financial losses estimated at €7 billion reflecting 16 million extra days of hospital stay. Each year 4 131 000 patients are affected by approximately 4 544 100 episodes of HAIs.

The total number of HAIs in European long-term care facilities (LTCFs) is estimated at 4.2 million per year.

8% to 12% of patients in developed countries is confronted with an adverse event (AE) during their hospital stay leading to (permanent) disability or even dead. As HAIs belong to one of the most important AEs they have a considerable economic impact prolonging hospital length of stay, increase readmission rates and necessitate additional ambulatory care or extra societal costs. The total preventable direct medical costs of AEs in the Netherlands are estimated as 1% of the national health care budget (94.2 billion 2013 - Statistics Netherlands).

Environmental cleanliness As antimicrobial resistance is a major and overall deteriorating public health problem international cooperation is necessary. Continued progress is needed to implement and improve programmes for the prevention and control of antimicrobial resistance and HAIs.

Environmental cleanliness might be one of the most important initiatives to reduce HAIs. Hospital surfaces are heavily contaminated with bacteria with the highest numbers on surfaces closest to the patients. Bed rails, nurse call buttons, curtains, towel dispensers, door handles, sinks, floors, clinical information stations, medical devices, stethoscopes, staff toilets etc. Actually, general hospital wards and Intensive Care Units are loaded with an abundance of potential pathogens. Surviving days, weeks or even months in the environment. Colonizing patients with bacteria from the hospital environment and getting HAIs or even die.

As most ventilator-associated pneumonias (VAPs) are the result of nosocomial microorganisms the environment plays an important role in the acquisition of pathogenic bacteria by contaminating health care workers hands and equipment. Furthermore, ICUs and wards struggle with colonized patients with ESBL-bacteria from sinks eventually leading to dead or outbreaks of group A streptococcus infections from contaminated curtains.

As key healthcare-associated pathogens have the capacity to persist for weeks to months on hospital surfaces indirect transmission is a serious threat, especially as antimicrobial resistance increases. Hospitalization in a room in which the previous patient had been colonized or infected with nosocomial pathogens (e.g. MRSA, VRE, multidrug-resistant Acinetobacter, Pseudomonas or C. difficile) has been shown to be a risk factor for colonization of infection with the same pathogen for the next patient. Furthermore, the most important risk factor for hand and glove contamination of healthcare workers with multidrug-resistant bacteria has been demonstrated to be positive environmental cultures. To decrease the frequency and level of contamination of environmental surfaces the Centre for Disease Control and Prevention recommends routine disinfection of medical equipment and environmental surfaces to prevent the spread of potential pathogens through the hospital ward or ICU. Improved room cleaning has shown to decrease the risk for MRSA, VRE and C. difficile acquisition. Unfortunately, environmental cleaning is frequently inadequate. Less than 50% of hospital room surfaces are adequately cleaned and disinfected even by environmental services personnel. Environmental services personnel have low wages, are under time pressure to clean rooms quickly with high turn-over rates of patients. Novel materials and cleaning technologies have been developed as ultraviolet germicidal irradiation (UVGI) or hydrogen peroxide vapor (HPV). However, both technologies are expensive and can just be used for terminal cleaning and not during routine daily care. Self-disinfecting surfaces may overcome these problems. Once applied antimicrobial surfaces will continuously reduce the bioburden of nosocomial pathogens preventing transmission and decrease HAIs.

MVX One of these self-disinfecting products is MVX. MVX contains titanium dioxide which by the use of nanotechnology is now available for use in the health sector. Working as a photocatalyticum it generates, in the presence of light, hydroxy radicals and oxygen radicals for at least five years after coating hospital surfaces (durability test TUV Rheinland). Laboratory tests show that MVX is effective in killing bacteria, viruses and fungi.

To the best of our knowledge there is just one study who examined the efficacy of titanium dioxide in reducing MRSA contamination in a hospital environment 19. In this cross-sectional observational study two ICU isolation rooms were coated and four beds in a 'Intermediate Care Area' (ICA). However, this study had some serious limitations. As 81% of all the samples (N=698) were taken from untreated surfaces there was a high chance of sampling bias. Especially as just 9% of all the samples were taken from the ICA, containing four of the six coated beds/rooms, against 48% of the ICU and 42% of a general ward. Furthermore, as just 10.6% of the samples were positive (N=74) we can really doubt about the validity of this study by the small sample size. Finally, countries with a low prevalence of MRSA (e.g. the Netherlands) are more interested in the prevalence of Enterobacteriaecae or non-MRSA (potential pathogenic microorganisms) and using a (semi)quantitative method.

This makes that the positive results reported on the effects of MVX from laboratory evaluations still have to be confirmed in the clinical setting. After getting the CE-marking Gelderse Vallei Hospital in Ede, the Netherlands, will be the first hospital in Europe to study the efficacy of MVX in the Intensive Care Unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the Intensive Care Unit and allocated to one of the four rooms

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Reduction in colony forming units cultured from T, S and E plates and culture sites taken in four week period after coating the rooms compared to amount of CFUs cultured from cultures and from culture sites taken in period before application MVX. | Up to 10 weeks
  Reduction in the total amount of all colony forming units (CFUs) cultured from all cultures (T, S and E plates) and from all culture sites taken in the four week period after coating of the rooms compared to the total amount of CFUs cultured from all cultures and from all culture sites taken in the period before application of MVX.

SECONDARY OUTCOMES:
Reduction in colony forming units cultured from T plates and from culture sites taken in four week period after coating the rooms compared to amount of CFUs cultured from T plates and from culture sites taken in the period before application of MVX. | Up to 10 weeks
Reduction in colony forming units cultured from S plates and from culture sites taken in four week period after coating the rooms compared to CFUs cultured from all S plates and from all culture sites taken in the period before application of MVX. | Up to 10 weeks
Reduction in colony forming units cultured from E plates and from culture sites taken in four week period after coating the rooms compared to the CFUs cultured from all E plates and from all culture sites taken in the period before application of MVX. | Up to 10 weeks
Number of positive microbiological culture plates (plates with ≥ 1 CFUs after 48 hrs of incubation) | Up to 10 weeks
Number of positive culture sites (plates of culture sites with ≥ 1 CFUs after 48 hrs of incubation) | Up to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arthur van Zanten, MD, PhD, Principal Investigator — Gelderse Vallei Hospital
Locations (1):
- Gelderse Vallei Hospital, Ede, Gelderland, Netherlands

REFERENCES:
- [Background] 2. European Centre for Disease Prevention and Control. Antimicrobial resistance surveillance in Europe 2012. Annual Report of the European Antimicrobial Resistance Surveillance Network (EARS-Net). Stockholm: ECDC; 2013.
- [Background] 3. www.who.int/gpsc/country_work/gpsc_ccisc_fact_sheet_en.pdf
- [Background] 4. European Centre for Disease Prevention and Control. Point prevalence survey of healthcare-associated infections and antimicrobial use in European long-term care facilities. April-May 2013. Stockholm: ECDC;2014.
- [Background] Zegers M, de Bruijne MC, Wagner C, Hoonhout LH, Waaijman R, Smits M, Hout FA, Zwaan L, Christiaans-Dingelhoff I, Timmermans DR, Groenewegen PP, van der Wal G. Adverse events and potentially preventable deaths in Dutch hospitals: results of a retrospective patient record review study. Qual Saf Health Care. 2009 Aug;18(4):297-302. doi: 10.1136/qshc.2007.025924. PMID 19651935
- [Background] Sousa P, Uva AS, Serranheira F, Nunes C, Leite ES. Estimating the incidence of adverse events in Portuguese hospitals: a contribution to improving quality and patient safety. BMC Health Serv Res. 2014 Jul 18;14:311. doi: 10.1186/1472-6963-14-311. PMID 25034870
- [Background] Hoonhout LH, de Bruijne MC, Wagner C, Zegers M, Waaijman R, Spreeuwenberg P, Asscheman H, van der Wal G, van Tulder MW. Direct medical costs of adverse events in Dutch hospitals. BMC Health Serv Res. 2009 Feb 9;9:27. doi: 10.1186/1472-6963-9-27. PMID 19203365
- [Background] Moore G, Muzslay M, Wilson AP. The type, level, and distribution of microorganisms within the ward environment: a zonal analysis of an intensive care unit and a gastrointestinal surgical ward. Infect Control Hosp Epidemiol. 2013 May;34(5):500-6. doi: 10.1086/670219. PMID 23571367
- [Background] Oberauner L, Zachow C, Lackner S, Hogenauer C, Smolle KH, Berg G. The ignored diversity: complex bacterial communities in intensive care units revealed by 16S pyrosequencing. Sci Rep. 2013;3:1413. doi: 10.1038/srep01413. PMID 23475210
- [Background] Shiferaw T, Beyene G, Kassa T, Sewunet T. Bacterial contamination, bacterial profile and antimicrobial susceptibility pattern of isolates from stethoscopes at Jimma University Specialized Hospital. Ann Clin Microbiol Antimicrob. 2013 Dec 13;12:39. doi: 10.1186/1476-0711-12-39. PMID 24330702
- [Background] Hota B. Contamination, disinfection, and cross-colonization: are hospital surfaces reservoirs for nosocomial infection? Clin Infect Dis. 2004 Oct 15;39(8):1182-9. doi: 10.1086/424667. Epub 2004 Sep 27. PMID 15486843
- [Background] Crnich CJ, Safdar N, Maki DG. The role of the intensive care unit environment in the pathogenesis and prevention of ventilator-associated pneumonia. Respir Care. 2005 Jun;50(6):813-36; discussion 836-8. PMID 15913471
- [Background] Joseph NM, Sistla S, Dutta TK, Badhe AS, Rasitha D, Parija SC. Role of intensive care unit environment and health-care workers in transmission of ventilator-associated pneumonia. J Infect Dev Ctries. 2010 Jun 3;4(5):282-91. doi: 10.3855/jidc.800. PMID 20539060
- [Background] Wolf I, Bergervoet PW, Sebens FW, van den Oever HL, Savelkoul PH, van der Zwet WC. The sink as a correctable source of extended-spectrum beta-lactamase contamination for patients in the intensive care unit. J Hosp Infect. 2014 Jun;87(2):126-30. doi: 10.1016/j.jhin.2014.02.013. Epub 2014 Apr 18. PMID 24831607
- [Background] Mahida N, Beal A, Trigg D, Vaughan N, Boswell T. Outbreak of invasive group A streptococcus infection: contaminated patient curtains and cross-infection on an ear, nose and throat ward. J Hosp Infect. 2014 Jul;87(3):141-4. doi: 10.1016/j.jhin.2014.04.007. Epub 2014 May 10. PMID 24928787
- [Background] 16. Steinberg et al. The role of the hospital environment in the prevention of healthcare-associated infections by contact transmission. HERD 2013;7(1):46-73.
- [Background] Weber DJ, Rutala WA. Understanding and preventing transmission of healthcare-associated pathogens due to the contaminated hospital environment. Infect Control Hosp Epidemiol. 2013 May;34(5):449-52. doi: 10.1086/670223. No abstract available. PMID 23571359
- [Background] 18. www.cdc.gov/hicpac/pdf/guidelines/disinfection_nov_2008.pdf
- [Background] 19. Leng et al. Efficacy of titanium dioxide compounds in preventing environmental contamination by meticillin resistant Staphylococcus aureus (MRSA). Int J Infect Control 2013, v9:i3.
- [Background] Shi H, Magaye R, Castranova V, Zhao J. Titanium dioxide nanoparticles: a review of current toxicological data. Part Fibre Toxicol. 2013 Apr 15;10:15. doi: 10.1186/1743-8977-10-15. PMID 23587290
- [Result] 1. European Centre for Disease Prevention and Control. Annual Epidemiological Report 2013. Reporting on 2011 surveillance data and 2012 epidemic intelligence data. Stockholm: ECDC; 2013.